CLINICAL TRIAL: NCT03200210
Title: Lowering-hyperuricemia Treatment on Cardiovascular Outcomes in Peritoneal Dialysis Patients: A Prospective, Multicenter, Double-Blinded, Randomized Controlled Trial
Brief Title: Lowering-hyperuricemia Treatment on Cardiovascular Outcomes in Peritoneal Dialysis Patients
Acronym: LUMINA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUMINA
Record Dates: First submitted 2017-06-25; First posted 2017-06-27 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hyperuricemia
Keywords: Continuous Ambulatory Peritoneal Dialysis (CAPD); Hyperuricemia; Cardiovascular events; Treatment
MeSH Terms: conditions — Hyperuricemia | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Febuxostat (Experimental): Febuxostat, starting at dose 20mg/d, once a day. And adjust dose according to serum uric acid at specific visits.
  Interventions: Drug: Febuxostat
- Treatment with placebo (Placebo Comparator): Same dose and dose adjustment as the intervention arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — Febuxostat tablets would be given to patients at dose of 20mg/d, once a day, and dose would be adjusted according to serum uric acid at specific visits.
  Other Names: Febuxostat Tablets
  Arms: Treatment with Febuxostat
Drug: Placebo — Pills manufactured to mimic Febuxostat tablets
  Arms: Treatment with placebo

SUMMARY:
The investigators will enroll continuous ambulatory peritoneal dialysis (CAPD) patients with hyperuricemia and randomly divide them into two groups, treated with Febuxostat and placebo respectively. After 3 years of following up, cardiovascular events, all cause mortality, cardiovascular mortality and non-fatal cardiovascular events are collected and recorded. The difference of cardiovascular events, all cause mortality and non-fatal cardiovascular event rate will be analyzed.

DETAILED DESCRIPTION:
The investigators anticipate enrolling 548 CAPD patients who have hyperuricemia in 21 centers and randomly allocate them into Febuxostat treatment group and placebo group. This study is double-blinded and will be followed up for 3 years. The primary endpoint is cardiovascular events, secondary endpoints are all-cause mortality, cardiovascular mortality and non-fatal cardiovascular events separately. All the endpoints will be collected, as well as other outcomes, such as blood pressure and dialysis dose and so on. The outcomes will be analyzed using statistics software.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects who are able to understand and have voluntarily signed the informed consent form (ICF)
* 18-70 years old at the time of randomization
* Subjects on PD for more than 3 months.
* Subjects have hyperuricemia, women: 6mg/dl(360μmol/L) <serum uric acid (sUA)<12mg/dl(720μmol/L); men: 7mg/dl(420μmol/L)<sUA<12mg/dl(720μmol/L).

Exclusion Criteria:

* 1.Subjects has history of gout
* Subjects who have a myocardial infarction, unstable angina,cardiovascular reconstructive surgery (such as a stent or bypass surgery), cerebrovascular accident 12 weeks prior to randomization, or plan cardiovascular reconstructive surgery during the trial
* Subjects who have New York stage IV heart failure occurs 4 weeks prior to the screening
* Subjects who have previously received renal transplantation and are currently prescribed immunosuppressive therapy
* Subjects who have severe liver disease, such as acute hepatitis, chronic active hepatitis, cirrhosis
* Subjects who have alanine aminotransferase (ALT) greater than 2 folds of the upper limited of normal or total bilirubin greater than 1.5 folds of upper limited of normal
* Subjects who have severe infections 4 weeks prior to the screening, such as pneumonia and peritoneal dialysis-related peritonitis;
* Subjects who have a major surgery 12 weeks prior to screening or not yet fully recovered from the surgery
* Subjects who have a malignancy
* Subjects who report a history of illicit drug use or a regular or daily alcohol consumption of≥4 alcoholic drinks per day in the 2 years before Screening
* Subjects who are allergic to Febuxostat
* Subjects who are enrolled in other clinical studies within 4 weeks or currently at randomization
* Subjects who are currently taking mercaptopurine, azathioprine, vidarabine, didanosine
* Subjects who are taking losartan, fenofibrate, thiazide diuretics or loop diuretics within 4 weeks at randomization
* Subjects who require long-term use of steroids (prednisone <30mg / d, or equivalent amount of other steroids and the use of <2 weeks can be enrolled)
* Subjects who require long-term use of salicylic acid drugs except low-dose aspirin
* Fertility, lactation patients unwilling or unable to contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 3 years
  Cardiovascular events compose of cardiovascular mortality and non-fatal cardiovascular events, cardiovascular mortality includes acute myocardial infarction, fatal arrhythmia, sudden death, cardiomyopathy, heart failure, and stroke; non-fatal cardiovascular events includes non-fatal acute myocardial infarction, hospital admission of heart failure, unstable angina, atherosclerotic disease needed hospitalization (including aneurysm, arterial dissection, arteriosclerosis occlusion), non-fatal stroke, transient ischaemic attack or lower limb ischaemia

SECONDARY OUTCOMES:
All-cause mortality | 3 years
  To record and calculate the deaths caused by any cause during follow up period
Cardiovascular mortality | 3 years
  To record and calculate the deaths cardiovascular mortality includes acute myocardial infarction, fatal arrhythmia, sudden death, cardiomyopathy, heart failure, and stroke during follow up period.
Non-fatal cardiovascular events | 3 years
  To record and calculate the non-fatal cardiovascular events including non-fatal acute myocardial infarction, hospital admission of heart failure, unstable angina, atherosclerotic disease needed hospitalization (including aneurysm, arterial dissection, arteriosclerosis occlusion), non-fatal stroke, transient ischaemic attack or lower limb ischaemia during follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen W, Huang N, Mao H, Yang X, Zhou Q, Jiang L, Ding J, Feng Q, Yu X. Rationale and design for Lowering-hyperUricaemia treatment on cardiovascular outcoMes In peritoNeal diAlysis patients: a prospective, multicentre, double-blind, randomised controlled trial (LUMINA). BMJ Open. 2020 Oct 10;10(10):e037842. doi: 10.1136/bmjopen-2020-037842. PMID 33040002